CLINICAL TRIAL: NCT03588195
Title: Evaluation of the Effectiveness of an Educational Program in Patients With Osteoarthritis of the Knee: a Randomized Controlled Trial
Brief Title: Educational Program for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Anamaria Jones, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP UNIFESP 458293
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Knee Osteoarthritis
Keywords: Education; Pain; Function; Quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental)
  Interventions: Other: Educational Program; Device: Transcutaneous Nerve Electro-Stimulation
- Control Group (Active Comparator)
  Interventions: Device: Transcutaneous Nerve Electro-Stimulation

INTERVENTIONS:
Other: Educational Program — Educational program consist in 5 consecutive sessions held once a week, with a duration of 60 minutes each class and at the end of the last class, a booklet was delivered for each patient with all the contents of the classes. This group also received Transcutaneous Nerve Electro-Stimulation twice weekly, for 5 weeks for 40 minutes each session
  Arms: Education Group
Device: Transcutaneous Nerve Electro-Stimulation — Transcutaneous Nerve Electro-Stimulation performed twice weekly, for 5 weeks for 40 minutes each session

SUMMARY:
Sixty patients with a diagnosis of knee osteoarthritis, aged between 40 and 80 years, of both genders were included. The patients were divided into: experimental group that carried out an educational program - 5 consecutive sessions held once a week, with a duration of 60 minutes each class and at the end of the last class, a booklet was delivered for each patient with all the contents of the classes and the Transcutaneous Nerve Electro-Stimulation device - being performed twice weekly, for 5 weeks for 40 minutes each session; and control group who only underwent treatment with the Transcutaneous Nerve Electro-Stimulation in the same parameters as experimental group. The evaluations were performed at the beginning of the treatment, 4 and 12 weeks after the beginning of the treatment using a numerical pain scale; WOMAC; IDATE and SF-36 questionnaires; and 6-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee Osteoarthritis by American College of Rheumatology criteria;
* Age between 40 and 80 years;
* Both genders;
* Numerical Pain Scale in the knee between 3 and 8 centimeters on a scale of 0 to 10 centimeters.

Exclusion Criteria:

* Systemic inflammatory diseases or any condition that prevents the practice of physical activity;
* Regular physical activity started or changed in the last twelve weeks;
* No ambulation;
* Joint injection in the knee in the previous twelve weeks;
* Previous knee surgery or surgery planned for the next twenty-four weeks;
* Physiotherapy in the last twelve weeks;
* Other disease that affects the lower limbs;
* Open wounds at the electrode application site;
* Planned trip in the next twelve weeks.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2018-06-17 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Baseline and after 4 and 12 weeks
  Evaluated using a numeric pain scale

SECONDARY OUTCOMES:
Change in function | Baseline and after 4 and 12 weeks
  Evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index
Change in Anxiety | Baseline and after 4 and 12 weeks
  Evaluated using the Inventory Anxiety Trait Inventory - State
Change in Generic Quality of life | Baseline and after 4 and 12 weeks
  Evaluated using the SF-36 questionnaire
Change in Functional capacity | Baseline and after 4 and 12 weeks
  Evaluated with the six minute walk test